CLINICAL TRIAL: NCT02756442
Title: Respiratory Disorder During Sleep in the Pregnancy : A Risk Factor in Gestational Diabetese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A01796-43; 2015-41 (Other: AP-HM)
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Disorder in Patient With Gestational Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregnant women with gestational diabetes (Experimental)
  Interventions: Other: Respiratory disorder assessment during sleep
- pregnant women without gestational diabetes (Active Comparator)
  Interventions: Other: Respiratory disorder assessment during sleep

INTERVENTIONS:
Other: Respiratory disorder assessment during sleep

SUMMARY:
Introduction:

The pregnancy brings about physiological and hormonal modifications which cause sleep disorder. The sleeplessness, snoring and a bad sleepquality are frequent during the pregnancy. Also a limited breathing airflow happens very often during the pregnancy. The limited airflow causes micro-awakenings that enter in the frame of the high resistances airways syndrome. To our knowledge there is no study about the outcome of micro-awakenings at pregnant women.

Objectives:

To compare the prevalence of the high resistances airways syndrome (RERA) in pregnant woman with or without gestational diabetes

Methods :

It is a monocentrical prospective study at pregnant women after the 30th amenorrhea week who consul the gynecologie and obstetrics department of the CHU NORD in Marseille. We are going to compare the breathing disorder during sleep of a control group with a group of women with gestational diabetes. A polysomnograph will be run at the included patients' home.

Expected results :

The physiological and hormonal modifications during the pregnancy could favor nocturnal sleep events (snoring, SAHOS and RERA) and its complications as gravidic HPN And gestational diabetes cause maternal and fœtal and morbidity and mortality. We put the hypothesis that limited airflow in association with micro-awakenings in the RERA have a negative impact on the glucose metabolism and favor the gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

Pregnant woman in the 3rd quarter of pregnancy (24 to 32 weeks amennorhea).

* Presenting a gestational diabetes ou not (=controle group)
* Written and signed consent.

Exclusion Criteria:

* Twin pregnancy
* High blood pressure before pregnancy
* Diabetes diagnosed before pregnancy
* Left ventricular ejection fraction below 40%
* Alcohol consumption (more than 7 glaces/day), drugs of type hypnotic, sedative, opioids
* History of gestational diabetes or glucose intolerance
* Severe cronical respiratory impairment (severe asthma)
* Creatinine clairance below 60 mL/min

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Respiratory Disturbance Index | 4 month
  Compare the respiratory disorder during sleep for pregnant women betwwen 2 groups with and without gestational diabetes based on RDI (Respiratory Disturbance Index)

SECONDARY OUTCOMES:
Air flow debit associated to micro awaking during sleep | 4 month
  To assess the resistance airways syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No